CLINICAL TRIAL: NCT04915430
Title: Comprehensive Supervised Heavy Training Program Versus Home Training Regimen in Patients With Subacromial Impingement Syndrome: a Randomized Trial.
Brief Title: Training in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reumatologiklinikken (Other)
Collaborators: Fonden for Faglig Udvikling af Speciallægepraksis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS_01
Record Dates: First submitted 2021-05-11; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Subacromial Impingement Syndrome
Keywords: shoulder; rotator cuff; exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients were randomized to either a supervised training regimen (STR) or a home training regimen
Who Masked: Investigator
Masking Description: The patients were blindly assigned to one of the training regimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised training regimen (Active Comparator): This training regimen consisted of 3 phases: the 1st focused on restoring motion, the 2nd on strengthening of the rotator cuff muscles, and the 3rd on strengthening of the scapular muscles. Stretching completed every training session.
  * Motion training consisted of 6 exercises.
    * Postural training: shoulder shrugs and shoulder retraction exercises.
    * Glenohumeral training: pendulum exercises, and active assisted flexion, abduction and external rotation.
  * Strengthening of the rotator cuff: side lying external rotation, internal rotation and scaption.
  * Strengthening of the scapular muscles: press-up, push-up with a plus, serratus anterior supine punch, standing rowing (low row), and seated rowing (high row).
  * Training sessions ended with 4 stretches: anterior shoulder stretch, posterior shoulder stretch, inferior capsular stretch, sleepers stretch.
  Exercises were performed 3 times a week, with progression after the 1st week, and thereafter every 2nd week.
  Interventions: Other: Training
- Home training regimen (Active Comparator): The program consisted of the following:
  * 1 motion exercise: upper trapezius relaxation
  * 3 strengthening exercises: serratus anterior strengthening exercise, humeral external rotation with the arm at the side of the body, and humeral external rotation with a rubber band and the arm at 90 degrees abduction.
  * 2 stretching exercises: posterior shoulder and pectoralis minor stretching, Exercises were performed daily, with weekly progression.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training

SUMMARY:
A randomized controlled trial comparing a comprehensive supervised training regimen with a validated home-based regimen for subacromial impingement syndrome.

DETAILED DESCRIPTION:
The purpose of the study is to compare a comprehensive supervised training regimen (STR) based on latest evidence including heavy slow resistance training with a validated home-based regimen (HTR). We hypothesized that the STR would be superior to the HTR.

Randomised control trial with blinded assessor. 126 consecutive patients with subacromial impingement syndrome were recruited and equally randomised to 12 weeks of either supervised training regimen (STR), or home-based training regimen (HTR). Primary outcomes were Constant Score (CS) and Shoulder Rating Questionnaire (SRQ) from baseline and 6 months after completed training. Results were analyzed according to intention-to treat principles.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial impingement syndrome

Exclusion Criteria:

* Ongoing claim with the Labour market insurance, insurance company or comparable institution.
* Ongoing application for job revalidation or health related pension.
* Radiating neck pain.
* Ultrasound verified complete rotator cuff tendon lesion, as defined by hypoechoic or anechoic full thickness defect of the tendon, or absence of the tendon.
* Periarthritis humeroscapularis.
* Acute luxation or fracture of the shoulder.
* Ongoing steady analgetic treatment of other concomitant painful condition, unrelated to the patients shoulder problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Shoulder constant score | 6 months after ended training
  Functional assessment of the shoulder
Shoulder Rating Questionnaire | 6 months after ended training
  Self-administered questionnaire

SECONDARY OUTCOMES:
Passive motion | 6 months after ended training
  Shoulder flexion, measurement in degrees; Shoulder abduction, measurement in degrees; Shoulder internal rotation, measurement in degrees; Shoulder external rotation, measurement in degrees.
Active motion | 6 months after ended training
  Shoulder flexion, measurement in degrees; Shoulder abduction, measurement in degrees; Shoulder internal rotation, measurement in degrees; Shoulder external rotation, measurement in degrees.
Visual Analogue Scale | 6 months after ended training
  Measurement of pain on a 10 cm scale, where 0 indicates no pain, and 10 worst pain for the following muscle tests: full can test, empty can test, lift off test, resisted external rotation, palm-up test, Yergason´s test.
Neer test | 6 months after ended training
  Stabilization of the patient's scapula with one hand, while passively flexing the arm while it is internally rotated. If the patient reports pain in this position, then the result of the test is considered to be positive (rated positive = 1 and negative = 0).
Hawkins test | 6 months after ended training
  Placing the patient's shoulder in 90 degrees of shoulder flexion with the elbow flexed to 90 degrees, and afterwards internally rotating the arm. The test is considered to be positive if the patient experiences pain with internal rotation (rated positive = 1 and negative = 0).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Schydlowsky, MD, PhD, Principal Investigator — Owner of the clinics

REFERENCES:
- [Derived] Schydlowsky P, Szkudlarek M, Madsen OR. Comprehensive supervised heavy training program versus home training regimen in patients with subacromial impingement syndrome: a randomized trial. BMC Musculoskelet Disord. 2022 Jan 15;23(1):52. doi: 10.1186/s12891-021-04969-0. PMID 35033043